CLINICAL TRIAL: NCT02167152
Title: Ischemic Preconditioning to Prevent Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00000718
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ischemic Preconditioning Group (Experimental): Participants randomized to this group will have a blood pressure cuff placed on each arm, and these cuffs will be inflated one at a time to a pressure calculated based on the person's blood pressure.
  Interventions: Other: Ischemic preconditionin
- Control Group (Active Comparator): Participants randomized to this group will have a blood pressure cuff placed on each arm, and these cuffs will be inflated one at a time to a set pressure (30mmHg, or millimeters of mercury on a blood pressure measuring machine).
  Interventions: Other: Ischemic preconditionin

INTERVENTIONS:
Other: Ischemic preconditionin — Ischemic preconditioning will be accomplished through 4 cycles of alternating 5-minute inflation and 5-minute deflation of an upper-arm blood pressure cuff to the patient's systolic blood pressure plus 50% to induce ischemia and reperfusion.

SUMMARY:
The purpose of this study is to learn about the impact of ischemic preconditioning in reducing contrast induced kidney damage in people with pre-existing kidney problems who are undergoing cardiac catheterization procedures.

DETAILED DESCRIPTION:
Ischemic preconditioning is thought to work by down-regulating pro-inflammatory gene expression and up-regulating anti-inflammatory gene expression in leukocytes. There is a local release of vasodilators, including adenosine and nitric oxide that are thought to have renal protective effects [16]. More is known regarding ischemic preconditioning in the heart, where it has been shown to decrease the adenine nucleotide pool, increase creatine phosphate and intracellular glucose, decrease ATP depletion, and lactate and H+ accumulation. This leads to sodium maintenance of the transmembrane sodium gradient that prevents intracellular edema. Ischemic preconditioning is thought to yield protection in the first minutes of reperfusion. Activation of the adenosine A1, bradykinin, and opioid receptors is thought to trigger protection. This is supported by the interference with protection if an adenosine receptor antagonist is administered. The role of reactive oxygen species as part of the protective mechanism has also been described via mitochondrial mKATP channels which lead to increased production of protective superoxide. Protein kinase C may also be involved in the protective mechanism of ischemic preconditioning, however the exact mechanism is unknown and controversial.

ELIGIBILITY:
Inclusion Criteria:

* Stage III-IV chronic kidney disease (with serum creatinine at or above 1.4 mg/dl and eGFR 15-55 ml/min/1.73m2 calculated by the Modification of Diet in Renal Disease formula)
* Undergoing planned coronary angiography (including both cardiac and peripheral vascular) and/or intervention at KUMC

Exclusion Criteria:

* Patients with normal renal function (stage 0 to 2 chronic kidney disease and/or serum creatinine less than 1.4 mg/dl)
* Inability or unwillingness to provide consent
* Patients undergoing hemodialysis or peritoneal dialysis therapy
* Patients with renal artery stenting
* Hemodynamically unstable patients
* Patients with acute or acute on chronic heart failure
* Patients who are unable to undergo the study procedure due to any upper extremity problems such as prior amputation, prior radical mastectomy, etc
* Patients who have not been hydrated prior to procedure using the standard protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 1 year
  Defined as an absolute increase in serum creatinine greater than or equal to 0.5 mg/dl or a relative increase of greater than or equal to 25% compared with pre-procedural baseline as compared to 48-72 hours post-angiography.

SECONDARY OUTCOMES:
Progression of kidney disease | 1 year
  Defined as change in serum creatinine and epidermal growth factor receptor (eGFR)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Gupta, MD, Principal Investigator — University of Kansas Medical Center; Patrick Tobbia, MD, Study Director — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States